CLINICAL TRIAL: NCT06587152
Title: Clinical Trial to Evaluate the Efficacy and Safety of Endoscopy System for General Surgery, Gynecology and Thoracic Surgery
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of a Thoracic and Abdominal Endoscopic Surgical System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cornerstone Robotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-00359-002
Record Dates: First submitted 2024-08-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pathologic Stage I Gastric Cancer AJCC v8; Colorectal Cancer; Esophageal Cancer; Hepatectomy; Radical Hysterectomy
Keywords: distal gastric cancer; radical surgery; colorectal cancer; oesophageal cancer; hepatectomy; radical hysterectomy
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted surgery (Experimental): Robot-assisted thoraco-laparoscopic esophagectomy
  Interventions: Procedure: Robot-assisted surgery

INTERVENTIONS:
Procedure: Robot-assisted surgery — Surgery with the Cornerstone Surgical Robot.

SUMMARY:
Evaluation of the efficacy and safety of thoracic and abdominal endoscopic surgical systems manufactured by Shenzhen Cornerstone Robotics Technology Co., Ltd. for use in general, gynaecological and thoracic surgical procedures.

DETAILED DESCRIPTION:
The trial was designed using a prospective, multi-centre, single-group target value approach.

For subjects who intend to undergo general surgery, gynaecological surgery and thoracic surgery assisted by the Thoracic and Abdominal Endoscopic Surgical System.

To use the Thoracic and Abdominal Endoscopic Surgical System developed by Shenzhen Cornerstone Robotics Technology Co., Ltd. to perform surgery in the above three disciplines, and to evaluate the efficacy and safety of the experimental medical device in the surgical treatment of the above three disciplines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years;
* Body Mass Height Index (BMI) 18<BMI<30kg/㎡;
* Patients identified by the investigator as suitable for general, gynaecological and thoracic surgery;
* Written informed consent.

Exclusion Criteria:

* Need for emergency surgery (e.g. gastric cancer, colorectal cancer combined with perforation, bleeding, obstruction, etc.);
* With other malignancies or a previous history of other malignancies.
* Preoperative imaging suggests that the tumour has distant metastases.
* The patient has a history of relevant surgery or previous history of other malignancy and is judged by the investigator to be unsuitable for enrolment.
* Severe bleeding tendencies or coagulopathic disorders.
* With long-term use of anticoagulant and anti-platelet drugs (anti-platelet aggregation drugs discontinued less than 1 week prior to surgery), history of bleeding disorders or hematopoietic or coagulation disorders.
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. systemic corticosteroids).
* Women who are pregnant or nursing an infant.
* With severe allergies and suspected or established alcohol, drug or substance addiction.
* Other conditions which, in the opinion of the investigator, make participation in this trial inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Surgical non-referral rate | during the surgery
  Surgical untransferred is defined as not converted from an experimental medical device assisted method to another surgical device control system assisted, laparoscopic surgery or open surgery.

SECONDARY OUTCOMES:
The surgeon's operating time | during the surgery
  Operative time（minutes）
Length of postoperative stay | up to 12 weeks
  Total number of days the patient was in hospital from the day of surgery to discharge.
Intraoperative blood loss | during the surgery
  Estimated blood loss（milliliters，ml）
Length of stay | The patient's total number of days from the day of surgery to discharge was recorded 30 days postoperatively.
  The postoperative day when patients complied with the predefined discharge criteria

CONTACTS AND LOCATIONS:
Overall Officials: Xiujun Cai, MD, Principal Investigator — President of Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine
Locations (1):
- Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JY, Ryu KW, Reim D, Eom BW, Yoon HM, Rho JY, Choi IJ, Kim YW. Robot-assisted gastrectomy for early gastric cancer: is it beneficial in viscerally obese patients compared to laparoscopic gastrectomy? World J Surg. 2015 Jul;39(7):1789-97. doi: 10.1007/s00268-015-2998-4. PMID 25670040
- [Background] Somashekhar SP, Deshpande AY, Ashwin KR, Gangasani R, Kumar R, Shetty S. Comparative Evaluation of the Short-Term Treatment Outcomes Between Open, Laparoscopic- and Robotic-Assisted Surgical Approaches for Rectal Cancer Treatment. Indian J Surg Oncol. 2020 Dec;11(4):649-652. doi: 10.1007/s13193-020-01137-z. Epub 2020 Jul 10. PMID 33299282
- See also: The adoption of robotic systems for gastric cancer surgery has been proven feasible and safe; however, a benefit over the laparoscopic approach has not yet been well-documented. — https://pubmed.ncbi.nlm.nih.gov/25670040/
- See also: The open surgeries and more recently minimal invasive surgeries aided by laparoscopic or robotic approaches are employed for rectal cancer treatment procedures. — https://pubmed.ncbi.nlm.nih.gov/33299282/